CLINICAL TRIAL: NCT06774937
Title: Clinical and Laboratory Profile of Myasthenia Gravis in Children At Sohag University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Menna Mohamed Sedik, Resident doctor of pediatric in ElHelal Hospital in Sohag, Sohag University
Other Study IDs: Soh-Med-24-09-03MS
Record Dates: First submitted 2024-12-11; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-06

CONDITIONS: Myasthenia Gravis in Children
MeSH Terms: interventions — Sex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- One group of patients againg one month to 16 years old with myasthenia gravis: Patients diagnosed with myasthenia gravis at the pediatric out patient clinic by clinical charactristics ,nerve study and laboratory data will be elligable for the study.
  Inclusion Criteria:
  * All patients from 1 month to 16 years confirmed diagnosis of myasthenia gravis by neurological and laboratory data.
  * Care giver accept to participate in the study.
  Interventions: Diagnostic Test: All patients in this study were subjected to the followings: (A) Clinical history focusing on: Sociodemographic data: age, gender , residence,and degree of consanguinity. Full neurodevelopmental his; Diagnostic Test: EMG ,rNST,Ach R antibodies & thyroid function

INTERVENTIONS:
Diagnostic Test: All patients in this study were subjected to the followings: (A) Clinical history focusing on: Sociodemographic data: age, gender , residence,and degree of consanguinity. Full neurodevelopmental his — Thorough clinical examination:
  1. General examination including general look, vital signs and anthropometric measurements.
  2. Scale system include gross motor function and muscle power(Quantitative Myasthenia Gravis Scale) [36] 3. detailed neurological examination including motor ,sensory and reflexes. (C) Investigations:
  1. Electrophysiological testing:
     EMG : is especially useful in diagnosis of seronegative MG and congenital myasthenic syndromes.
     NCS: including repetitive nerve stimulation test (r NST)
  2. laboratory studies:
     * Serology. Detection of antibodies to the AChR supports the diagnosis of JMG. In young children where AChR antibodies are negative this can lead to difficulty in differentiating from CMS.
     * Thyroid function tests :
  3. Imaging:
     • CT chest: Although thymoma in children is rare, the thymus must be imaged once JMG has been diagnosed.
  4. molecular studies (when possible).
Diagnostic Test: EMG ,rNST,Ach R antibodies & thyroid function — C) Investigations:
  1. Electrophysiological testing:
     EMG : is especially useful in diagnosis of seronegative MG and congenital myasthenic syndromes.
     NCS: including repetitive nerve stimulation test (r NST)
  2. laboratory studies:
     * Serology. Detection of antibodies to the AChR supports the diagnosis of JMG. In young children where AChR antibodies are negative this can lead to difficulty in differentiating from CMS.
     * Thyroid function tests :
  3. Imaging:
     • CT chest: Although thymoma in children is rare, the thymus must be imaged once JMG has been diagnosed.
  4. molecular studies (when possible).

SUMMARY:
This study includes clinical and laboratory studies of patients with Myathenia gravis at Sohag Neurology outpatient clinic of pediatric department

DETAILED DESCRIPTION:
All patients in this study were subjected to the followings:

(A) Clinical history focusing on: Sociodemographic data: age, gender , residence,and degree of consanguinity. Full neurodevelopmental history: neurological evaluation Family history. Mode of delivery

(B) Thorough clinical examination: General examination including general look, vital signs and anthropometric measurements.

Scale system include gross motor function and muscle power(Quantitative Myasthenia Gravis Scale) [36] detailed neurological examination including motor ,sensory and reflexes. (C) Investigations:

1. Electrophysiological testing:

   EMG : is especially useful in diagnosis of seronegative MG and congenital myasthenic syndromes.

   NCS: including repetitive nerve stimulation test (r NST)
2. laboratory studies: Serology. Detection of antibodies to the AChR supports the diagnosis of JMG. In young children where AChR antibodies are negative this can lead to difficulty in differentiating from CMS.

   Thyroid function tests :
3. Imaging:

   CT chest: Although thymoma in children is rare, the thymus must be imaged once JMG has been diagnosed.
4. molecular studies (when possible).

ELIGIBILITY:
Inclusion Criteria:

* All patients from 1 month to 16 years confirmed diagnosis of myasthenia gravis by neurological and laboratory data.

Care giver accept to participate in the study.

Exclusion Criteria:

* Failure to obtain informed consent. Other neurological and neuromuscular disorders. Age above 16 years.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients:
  Patients diagnosed with myasthenia gravis at the pediatric out patient clinic by clinical charactristics ,nerve study and laboratory data will be elligable for the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and laboratory profile of patients with myasthenia gravis at Sohag Neurology Outpatient clinic of pediatric department | Follow up for 6 months
  All patients with myasthenia gravis in this study focusing on clinical and laboratory profile at Sohag Neurology outpatient clinic.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag University Hospital, Sohag, Sohag Governorate
  - Sohag university, Sohag

IPD SHARING:
Plan to Share IPD: Undecided